CLINICAL TRIAL: NCT00818935
Title: Glycemic Indices of Caribbean Foods and Application in Dietary Lifestyle Intervention for Management of Type 2 Diabetes Mellitus
Brief Title: Low-Intermediate-Glycemic Index Caribbean Foods Versus High Glycemic Index Foods in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of the West Indies (Other)
Responsible Party: Dr. Andrew Wheatley (Principal Investigator), University of the West Indies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWI-0012
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes; Inflammation; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-Intermediate-Glycemic Index diets (Experimental)
  Interventions: Dietary Supplement: Low-Intermediate-Glycemic Index diets
- High GI diet (Active Comparator)
  Interventions: Dietary Supplement: High GI diet

INTERVENTIONS:
Dietary Supplement: Low-Intermediate-Glycemic Index diets
  Arms: Low-Intermediate-Glycemic Index diets
Dietary Supplement: High GI diet
  Arms: High GI diet

SUMMARY:
The purpose of this study is to determine whether low and intermediate GI Caribbean foods are effective in the management of type 2 diabetes.

DETAILED DESCRIPTION:
Recruitment: Subjects for the study were sourced primarily from the University Hospital of the West Indices (Diabetic Clinic) and from the Diabetes Association of Jamaica Outreach Centers in Kingston and St. Catherine. Volunteers were also recruited through clinical visits and by opportunistic population screenings and by placing advertisements in local newspapers and by distributing similar advertisements to the diabetes clinic and diabetes education programs.

Information Sessions: Approximately 112 volunteers in groups of 10-30 with or without spouses will attend one of a number of evening information sessions at run from the Department of Basic Medical Sciences (Biochemistry Section), University of the West Indies. During the sessions the exact nature of the study will be described and volunteers will have the opportunity to ask specific questions about the study.

Screening: Potential subjects will then fill in and return to the investigators a detailed questionnaire concerning their medical history, medications (including vitamin, mineral and nutritional supplements) smoking habits, alcohol intake and exercise pattern and whether they are currently on a specific diet. Details will also be obtained concerning planned vacations. Those subjects deemed potentially eligible will be asked to give a fasting blood sample at the Biotechnology Center, University of the West Indies. Individuals who meet the study criteria, are invited to return again to the Department. The principles of the diabetic diet which they are already expected to be following will be reinforced by the study nutritionist whereby consuming a diet with more than 50% of daily calories from carbohydrate; less than 10% from saturated fat and 20% from mono- and polyunsaturated fat, or up to 25% if the surplus is from monounsaturated fat; cholesterol less than 300 mg/day; and approximately 1.0 g protein per kg ideal weight per day. An increase in the intake of dietary fiber to 15 g per 1000 kcal was encouraged. All subjects were then randomized to one 24-week treatment in a two-treatment parallel design.

Treatments: 1) low glycemic index dietary advice (e.g. to eat intact grain cereals, boiled green banana, boiled sweet potato, boiled round leaf yellow yams and boiled breadfruit) 2) high cereal fiber diet. Background diets will be the subjects' diabetic diets, modified as above, which will conform. Diet histories will be recorded at weekly for 24 weeks. These diets will be assessed for consistency by the dietitian in the subject's presence through dietary recall and semi-quantitative assessment of food portion sizes consumed. Where necessary, modifications in diet will be made to ensure weight maintenance. Compliance will be assessed by 7 day food records.

Duration: the study will consist of four months recruitment and patient selection, during which time estimation of individual caloric requirements will be performed, and 6 months treatment period.

Study Details: Fasting blood samples were obtained at day zero and weeks 2, 4, 8, 12, 16 and 24 of each study period. Twenty-four hour urine for urinary C-peptide analyses will be obtained immediately prior to the beginning of the study and at the end of each 24-week treatment phase.

Palatability and satiety: subjects will record their ratings using a 9-point bipolar semantic scale at weekly intervals during each study phase.

Anthropometric measures: height at recruitment, waist and hip circumference, and body composition will be taken immediately prior to and at the end of each study phase. Body weight and blood pressure will be measured at clinic visits.

This study will help to indicate whether a low-intermediate-GI indigenous Caribbean foods dietary advice can reduce the postprandial glycemia, inflammation and cardiovascular risks in person with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* between the age group of 25-65 years who have been previously clinically diagnosed with type 2 diabetes mellitus.
* Subjects were required to have low activity jobs, for example, clerical jobs

Exclusion Criteria:

* Individuals with Impaired glucose tolerance (IGT)
* Diabetics who were treated with insulin
* Subjects who were on hypertensive medications
* Individuals who are polycythemic or anemic
* Type 2 diabetics who participate in vigorous exercise Persons with chronic disease other than diabetes making a 3-year survival improbable as well as other medical characteristics that are likely to interfere with their participation in the study, for example, subjects with unbalanced clinical conditions, such as thyroid and liver disease, which could interfere with glucose metabolism; alcoholism or inability to effectively participate in a dietary programme

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Glycated Haemoglobin | 6 months

SECONDARY OUTCOMES:
body weight, homocysteine, C-reactive protein, plasma lipids and lipoproteins, fasting body glucose, insulin, insulin resistance, serum urea, creatinine, C-peptide | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Helen N Asemota, PhD, Principal Investigator — Univeristy of the West Indies
Locations (1):
- University of the West Indies, Kingston, Jamaica